CLINICAL TRIAL: NCT03365089
Title: Prospective Randomized Evaluation of the Effect of Ligation of Venous Side Branches in Dialysis Arteriovenous Fistulas Presenting With Failure to Mature
Brief Title: Collateral Ligation in Failing Fistulas
Acronym: CLiFF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Zubin Irani, Instructor in Inteventional Radiology, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017P001237
Record Dates: First submitted 2017-11-21; First posted 2017-12-07 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Hemodialysis Access Failure
Keywords: Hemodialysis fistula; Failure to mature; Collateral vein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collateral vein ligation (Experimental): Ligation of collateral veins under sonographic guidance
  Interventions: Procedure: Collateral vein ligation
- Control (No Intervention): No collateral vein ligation.

INTERVENTIONS:
Procedure: Collateral vein ligation — Collateral venous flow will be interrupted by ultrasound-guided ligation of venous side branches.
  Arms: Collateral vein ligation

SUMMARY:
Arteriovenous fistulas (AVFs) for hemodialysis often fail to become usable due to failure to mature (FTM). The most common cause is narrowing of the artery or vein (stenosis). Another potential cause is the presence of collateral or side branch veins that steal blood flow from the main fistula channel. Some believe that occluding these veins might help maturation of those failing AVFs. To evaluate if this actually works, patients with FTM will be randomly assigned to side branch vein ligation (or not), and rates of AVF maturation of the two groups will be compared.

DETAILED DESCRIPTION:
Arteriovenous fistulas (AVFs) for hemodialysis often fail to become usable due to failure to mature (FTM). The most common cause is stenosis of the artery or vein. Another potential cause is the presence of collateral or side branch veins that steal blood flow from the main fistula channel. The utility of ligating these veins to improve maturation of those failing AVFs is controversial. To evaluate this, 35 patients presenting for fistulograms for evaluation of AVFs with FTM, found to have side branch veins will be prospectively enrolled. After management of stenoses (if present), they will be randomly assigned to ligation of the venous side branches or not. Maturation rates for each group will be prospectively assessed. For patients assigned to the control group who have persistent failure to mature, a cross-over intervention will be performed and side branch ligation will be offered.

ELIGIBILITY:
Inclusion criteria:

- Patients with upper extremity autogenous AVF presenting with FTM with evidence of collaterals on ultrasound and/or clinical exam.

Exclusion criteria:

* Age under 18 years
* Pregnant women
* Prior endovascular or surgical procedure in the fistula after its creation (with the exception of surgical superficialization or mobilization)
* Clinical evidence of infection associated with the AVF
* Uncorrectable coagulopathy (International Normalized Radio >2.5, platelet count <50.000/μL)
* Absence of significant venous side branches on angiogram (defined as those that arise in the initial 10 cm, including the future cannulation zone, and have maximal diameter greater than or equal to one third of the widest diameter of the fistula's main venous channel in this segment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Fistula maturation rate | 8 weeks after randomization
  Proportion of patients with usable arteriovenous fistula at the end of the study (being able to deliver the prescribed dialysis dose 75% of the sessions in the first 4 weeks of use via 2 needles)

CONTACTS AND LOCATIONS:
Overall Officials: Zubin Irani, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sidawy AN, Spergel LM, Besarab A, Allon M, Jennings WC, Padberg FT Jr, Murad MH, Montori VM, O'Hare AM, Calligaro KD, Macsata RA, Lumsden AB, Ascher E; Society for Vascular Surgery. The Society for Vascular Surgery: clinical practice guidelines for the surgical placement and maintenance of arteriovenous hemodialysis access. J Vasc Surg. 2008 Nov;48(5 Suppl):2S-25S. doi: 10.1016/j.jvs.2008.08.042. PMID 19000589
- [Background] Lok CE. Fistula first initiative: advantages and pitfalls. Clin J Am Soc Nephrol. 2007 Sep;2(5):1043-53. doi: 10.2215/CJN.01080307. Epub 2007 Aug 16. No abstract available. PMID 17702726
- [Background] Patel ST, Hughes J, Mills JL Sr. Failure of arteriovenous fistula maturation: an unintended consequence of exceeding dialysis outcome quality Initiative guidelines for hemodialysis access. J Vasc Surg. 2003 Sep;38(3):439-45; discussion 445. doi: 10.1016/s0741-5214(03)00732-8. PMID 12947249
- [Background] Miller PE, Tolwani A, Luscy CP, Deierhoi MH, Bailey R, Redden DT, Allon M. Predictors of adequacy of arteriovenous fistulas in hemodialysis patients. Kidney Int. 1999 Jul;56(1):275-80. doi: 10.1046/j.1523-1755.1999.00515.x. PMID 10411703
- [Background] Lok CE, Oliver MJ, Su J, Bhola C, Hannigan N, Jassal SV. Arteriovenous fistula outcomes in the era of the elderly dialysis population. Kidney Int. 2005 Jun;67(6):2462-9. doi: 10.1111/j.1523-1755.2005.00355.x. PMID 15882293
- [Background] Dixon BS, Novak L, Fangman J. Hemodialysis vascular access survival: upper-arm native arteriovenous fistula. Am J Kidney Dis. 2002 Jan;39(1):92-101. doi: 10.1053/ajkd.2002.29886. PMID 11774107
- [Background] Miller CD, Robbin ML, Allon M. Gender differences in outcomes of arteriovenous fistulas in hemodialysis patients. Kidney Int. 2003 Jan;63(1):346-52. doi: 10.1046/j.1523-1755.2003.00740.x. PMID 12472802
- [Background] Allon M, Robbin ML. Increasing arteriovenous fistulas in hemodialysis patients: problems and solutions. Kidney Int. 2002 Oct;62(4):1109-24. doi: 10.1111/j.1523-1755.2002.kid551.x. PMID 12234281
- [Background] Sidawy AN, Gray R, Besarab A, Henry M, Ascher E, Silva M Jr, Miller A, Scher L, Trerotola S, Gregory RT, Rutherford RB, Kent KC. Recommended standards for reports dealing with arteriovenous hemodialysis accesses. J Vasc Surg. 2002 Mar;35(3):603-10. doi: 10.1067/mva.2002.122025. PMID 11877717
- [Background] Dariushnia SR, Walker TG, Silberzweig JE, Annamalai G, Krishnamurthy V, Mitchell JW, Swan TL, Wojak JC, Nikolic B, Midia M; Society of Interventional Radiology Standards of Practice Committee. Quality Improvement Guidelines for Percutaneous Image-Guided Management of the Thrombosed or Dysfunctional Dialysis Circuit. J Vasc Interv Radiol. 2016 Oct;27(10):1518-30. doi: 10.1016/j.jvir.2016.07.015. Epub 2016 Sep 9. No abstract available. PMID 27622727
- [Background] Nassar GM. Endovascular management of the "failing to mature" arteriovenous fistula. Tech Vasc Interv Radiol. 2008 Sep;11(3):175-80. doi: 10.1053/j.tvir.2008.09.004. PMID 19100946
- [Background] Beathard GA, Settle SM, Shields MW. Salvage of the nonfunctioning arteriovenous fistula. Am J Kidney Dis. 1999 May;33(5):910-6. doi: 10.1016/s0272-6386(99)70425-7. PMID 10213648
- [Background] Han M, Kim JD, Bae JI, Lee JH, Oh CK, Ahn C, Won JH. Endovascular treatment for immature autogenous arteriovenous fistula. Clin Radiol. 2013 Jun;68(6):e309-15. doi: 10.1016/j.crad.2013.01.005. Epub 2013 Mar 5. PMID 23465323
- [Background] Ahmed O, Patel M, Ginsburg M, Jilani D, Funaki B. Effectiveness of collateral vein embolization for salvage of immature native arteriovenous fistulas. J Vasc Interv Radiol. 2014 Dec;25(12):1890-4. doi: 10.1016/j.jvir.2014.08.015. Epub 2014 Oct 3. PMID 25280664
- [Background] Cui J, Freed R, Liu F, Irani Z. Interrupting Rivaling Access-flow with Nonsurgical Image-guided ligation: the "IRANI" Procedure. Semin Dial. 2015 Nov-Dec;28(6):E53-7. doi: 10.1111/sdi.12450. PMID 26507374
- [Background] Turmel-Rodrigues LA. Mechanical enhancement of AVF maturation. J Vasc Access. 2014;15 Suppl 7:S55-9. doi: 10.5301/jva.5000232. Epub 2014 Apr 12. PMID 24817456
- [Background] Haq NU, Albaqumi M. Accessory vein obliteration criteria for immature fistulae: a modest proposal for an old paradigm. Semin Dial. 2014 Sep-Oct;27(5):E51-4. doi: 10.1111/sdi.12239. Epub 2014 May 6. PMID 24796386
- See also: Fistula First National Vascular Access Improvements Initiative — https://www.esrdncc.org/en/fistula-first-catheter-last